CLINICAL TRIAL: NCT01608113
Title: Long-term Follow-up of Subfoveal Neovascular AMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christopher Kiss, Head of Vienna Study Center, Medical University of Vienna
Other Study IDs: EK 802/2011
Record Dates: First submitted 2012-04-10; First posted 2012-05-30 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2012-05

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: neovascular AMD; Optical coherence tomography; reading acuity; contrast sensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Treatment naive patients with subfoveal nAMD initially treated monthly with intravitreal anti-VEGF and subsequently PRN, will be included in this study. Patients will be investigated for the first 2 years monthly and subsequently according to disease activity but at least every two months. Patients will be examined with 4m BCVA ETDRS distance visual acuity, reading acuity measured by Radner-Reading-Charts, contrast sensitivity by Pelli-Robson score, microperimetry and HD-OCT.

ELIGIBILITY:
Inclusion Criteria:

* treatment naive subfoveal AMD, written informed consent, able to read

Exclusion Criteria:

* choroidal neovascularisation due to other ocular diseases, mature cataract

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering on treatment naive subfoveal neovascular age-related macular degeneration
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2011-09

PRIMARY OUTCOMES:
Long-term visual function performance | four years

SECONDARY OUTCOMES:
change of morphological alterations assessed by SD-OCT | four years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Kiss, MD, Principal Investigator — Medical University Vienna
Locations (1):
- Department of Ophthalmology Medical University of Vienna, Vienna, Vienna, Austria